CLINICAL TRIAL: NCT06957093
Title: Evaluation of the Therapeutic Efficacy and Safety of Artificial Intelligence-based Decision-making Technology in the Integrated Management of Diabetes Mellitus: a Longitudinal, Open-labeled, Randomized Controlled Trial
Brief Title: Therapeutic Efficacy and Safety Evaluation of AI in the Management of Diabetes: A RCT Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K2024283
Record Dates: First submitted 2025-04-17; First posted 2025-05-04 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus Type 2 (T2DM); Artificial Intelligence (AI)
Keywords: Diabetes mellitus type 2 (T2DM); Artificial Intelligence (AI)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Artificial Intelligence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artificial Intelligence Intervention Group (Experimental): The patients will be trained to independently use the diabetes telemedicine platform application. Each patient will be equipped with a glucometer and exercise bracelet, and the data will be automatically transmitted to the medical server via Bluetooth. The healthcare platform will analyze the uploaded data and provide feedback suggestions on medication, diet, and exercise automatically. The platform will also monitor the medical and lifestyle data of the patients every two weeks,offer feedback based on the analyses, and remind the patient to adhere to the self-management protocol based on the platform. Free outpatient visits will be provided to both the intervention and control groups every twelve weeks.
  Interventions: Other: artificial intelligence
- Conventional Treatment Group (Active Comparator): Patients in the control group will receive a free blood glucometer and will have regular outpatient appointments every 12 weeks..
  Interventions: Other: Routine diagnosis and treatment group for diabetes

INTERVENTIONS:
Other: artificial intelligence — The platform will also monitor the medical and lifestyle data of the patients every two weeks,offer feedback based on the analyses, and remind the patient to adhere to the self-management protocol based on the platform.
  Arms: Artificial Intelligence Intervention Group
Other: Routine diagnosis and treatment group for diabetes — There is no limit to the number of outpatient visits for the control group; however, they are required to regularly monitor and record their blood glucose, diet, and exercise data to ensure that the medical team (endocrinologist and nutritionist) objectively conducttheir diagnosis and treatment activities. The medical team will provide free outpatient visits every 12 weeks, along with advice on medication, diet, and exercise based on the individual's blood glucose level.
  Arms: Conventional Treatment Group

SUMMARY:
Purpose: To evaluate the efficacy of artificial intelligence (AI)-based decision-making technology in managing glycated hemoglobin (HbA1c) and blood glucose levels compared to the control group.

Methods: For the AI Intervention group, the patients will be trained to independently use the diabetes telemedicine platform application. Each patient will be equipped with a glucometer and exercise bracelet, and the data will be automatically transmitted to the medical server via Bluetooth. The healthcare platform will analyze the uploaded data and provide feedback suggestions on medication, diet, and exercise automatically. The platform will also monitor the medical and lifestyle data of the patients every two weeks, offer feedback based on the analyses, and remind the patient to adhere to the self-management protocol based on the platform. The platform is a digitally integrated healthcare platform that patients can use independently without the need for monitoring and assistance by healthcare professionals. The glucometer and pedometer bracelet will automatically connect to the platform through Bluetooth. The patient lab sheet identification and structured conversion system, AI for food picture identification and calorie calculation systems, and the AI decision-making system are on the cloud server. Patients upload image information, such as lab sheets and meal pictures, through the patient's diabetes mobile health system, and the cloud platform intelligently analyzes the patient's disease, medication, and daily life status to develop personalized solutions according to individual control goals. Free outpatient visits will be provided to both the intervention and control groups every twelve weeks. For the conventional treatment group, patients will receive a free blood glucometer and will have regular outpatient appointments. There is no limit to the number of outpatient visits; however, they are required to regularly monitor and record their blood glucose, diet, and exercise data to ensure that the medical team objectively conduct their diagnosis and treatment activities. The medical team will provide free outpatient visits every 12 weeks, along with advice on medication, diet, and exercise based on the individual's blood glucose level.

Expected results: A significant difference in HbA1c change from baseline to 48 weeks and improved FPG and 2-hour postprandial blood glucose levels in the AI intervention group were observed.

DETAILED DESCRIPTION:
Follow-up Plan::

Visit 1(-4W~-1W): Obtain the written informed consents of the patients, conduct the demographic survey, medical record survey, drug history investigation, subject compliance investigation, vital signs checkup, laboratory tests, imaging, and other instrument examinations, as well as evaluate the comorbidities of diabetes.

Visit 2 (D0): Educate the intervention group operating the platform system, evaluating diabetic hypoglycemia events, enhancing patients' self-management abilities, and knowledge mastery. Lab tests will be conducted at 12-week intervals, including Visit 3 (12W), Visit 4 (24W) or Visit 5 (36W), and Visit 6 (48W).

ELIGIBILITY:
Inclusion Criteria：

* Age: ≥18 years，≤75 years;
* Diagnosed with type 2 diabetes for ≥1 year;
* 7.0% ≤HbA1c ≤11%;
* Body mass index ≥18.5 kg/m2;
* Proficient ability to use smart phones;
* Agreed to utilize a digital integrated healthcare platform for diabetes care and research;
* Informed consents are obtained from the participants.

Exclusion Criteria:

* Presence of other types of diabetes, such as type 1 diabetes and gestational diabetes;
* Severe diabetic complications;
* Medical history of chronic liver diseases, including hemochromatosis, hepatocellular carcinoma, autoimmune liver disease, cirrhosis, viral hepatitis (including hepatitis A, B, and C), or hepatolenticular degeneration;
* Kidney injury (serum creatinine ≥1.5 times the upper limit of the reference) ; Serum ALT and AST levels elevated >2-fold;
* Medical history of mental disorders, such asschizophrenia, depression, or bipolar affective disorder;
* Excessive alcohol intake or drug abuse in the past 3 months;
* Use of medications affecting glucose metabolism, such as corticosteroids or ·consumption of immunosuppressive and anti-obesity medications in the past 3 months;
* Pregnancy, planning for pregnancy, or lactation; or any other conditions unsuitable for trial participation;
* Participatingor plan to participate in other clinical trials; and other cases that are inappropriate to participate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 48weeks
  Change From Baseline in HbA1c levels at 24 and 48 Weeks
Fasting Blood Glucose (FBG) | 48 weeks
  Change from baseline in mean fasting blood glucose at 48 weeks
2-hour Postprandial Blood Glucose (2hPPG) | 48 weeks
  Change from baseline in mean 2-hour postprandial blood glucose at 48 weeks
Hypoglycemic events | 48 weeks
  Number of hypoglycemic events from baseline to 48 weeks

SECONDARY OUTCOMES:
Healthcare expenses | 48weeks
  Assess the monthly treatment costs from baseline to the 48 weeks
Insulin and oral hypoglycemic agent dosing | 48 weeks
  Changes in oral medication and insulin dosage from baseline to week 48
Serum lipids | 48 weeks
  Change From Baseline in serum lipids levels at 48 Weeks
blood pressure | 48 weeks
  Change From Baseline in blood pressure at 48 Weeks
BMI | 48 weeks
  Weight in kilograms, height in meters, weight and height will be combined to report BMI in kg/m^²
body weight | 48weeks
  weight in kilograms
Fasting C-peptide level | 48weeks
  Change From Baseline in fasting C-peptide level at 6 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chenglin Sun, Doctor, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee YB, Kim G, Jun JE, Park H, Lee WJ, Hwang YC, Kim JH. An Integrated Digital Health Care Platform for Diabetes Management With AI-Based Dietary Management: 48-Week Results From a Randomized Controlled Trial. Diabetes Care. 2023 May 1;46(5):959-966. doi: 10.2337/dc22-1929. PMID 36821833
- [Background] Kim EK, Kwak SH, Jung HS, Koo BK, Moon MK, Lim S, Jang HC, Park KS, Cho YM. The Effect of a Smartphone-Based, Patient-Centered Diabetes Care System in Patients With Type 2 Diabetes: A Randomized, Controlled Trial for 24 Weeks. Diabetes Care. 2019 Jan;42(1):3-9. doi: 10.2337/dc17-2197. Epub 2018 Oct 30. PMID 30377185
- [Background] Dobson R, Whittaker R, Jiang Y, Maddison R, Shepherd M, McNamara C, Cutfield R, Khanolkar M, Murphy R. Effectiveness of text message based, diabetes self management support programme (SMS4BG): two arm, parallel randomised controlled trial. BMJ. 2018 May 17;361:k1959. doi: 10.1136/bmj.k1959. PMID 29773539
- [Background] Agarwal P, Mukerji G, Desveaux L, Ivers NM, Bhattacharyya O, Hensel JM, Shaw J, Bouck Z, Jamieson T, Onabajo N, Cooper M, Marani H, Jeffs L, Bhatia RS. Mobile App for Improved Self-Management of Type 2 Diabetes: Multicenter Pragmatic Randomized Controlled Trial. JMIR Mhealth Uhealth. 2019 Jan 10;7(1):e10321. doi: 10.2196/10321. PMID 30632972
- [Background] Doupis J, Festas G, Tsilivigos C, Efthymiou V, Kokkinos A. Smartphone-Based Technology in Diabetes Management. Diabetes Ther. 2020 Mar;11(3):607-619. doi: 10.1007/s13300-020-00768-3. Epub 2020 Jan 25. PMID 31983028
- [Background] Sun C, Sun L, Xi S, Zhang H, Wang H, Feng Y, Deng Y, Wang H, Xiao X, Wang G, Gao Y, Wang G. Mobile Phone-Based Telemedicine Practice in Older Chinese Patients with Type 2 Diabetes Mellitus: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2019 Jan 4;7(1):e10664. doi: 10.2196/10664. PMID 30609983
- [Background] Wang H, Yuan X, Wang J, Sun C, Wang G. Telemedicine maybe an effective solution for management of chronic disease during the COVID-19 epidemic. Prim Health Care Res Dev. 2021 Sep 29;22:e48. doi: 10.1017/S1463423621000517. PMID 34583801
- [Background] Bulut C, Kato Y. Epidemiology of COVID-19. Turk J Med Sci. 2020 Apr 21;50(SI-1):563-570. doi: 10.3906/sag-2004-172. PMID 32299206
- [Background] Mahajan V, Singh T, Azad C. Using Telemedicine During the COVID-19 Pandemic. Indian Pediatr. 2020 Jul 15;57(7):652-657. Epub 2020 May 14. PMID 32412914